CLINICAL TRIAL: NCT01583322
Title: Randomized Double Blind Placebo-controlled Phase II Trial of Vargatef® (Nintedanib) in Addition to First Line Chemotherapy With Interval Debulking Surgery in Patients With Adenocarcinoma of the Ovary, the Fallopian Tube or Serous Adenocarcinoma of the Peritoneum
Brief Title: Vargatef in Addition to First Line Chemotherapy With Interval Debulking Surgery in Patients With Ovarian Cancer
Acronym: CHIVA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ARCAGY/ GINECO GROUP (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GINECO-OV119
Record Dates: First submitted 2012-04-19; First posted 2012-04-24 (Estimated); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Ovarian Cancer
Keywords: ovarian cancer; debulking surgery; interval debulking; vargatef; nintedanib; maintenance; first line; paclitaxel; carboplatin
MeSH Terms: conditions — Ovarian Neoplasms | interventions — nintedanib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vargatef/Nintedanib (Experimental)
  Interventions: Drug: vargatef
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: vargatef — 400 mg (200 mg twice daily) Route of administration= oral Twice daily (to be swallowed unchewed with a glass of water of about 250 mL. If taken twice the dose interval should be of around 12 hours at the same times every day, usually in the morning and the evening after food intake).
  Continuous daily dosing until progression of disease or until criteria for interruption of treatment are met, no intake of Vargatef® (Nintedanib) on days of paclitaxel and carboplatin administration. The maximum time on monotherapy is 2 years.
  Arms: vargatef/Nintedanib
Drug: placebo — Contains 0 mg of Vargatef® (Nintedanib) in capsules matching 100 mg and 150 mg of Vargatef® (Nintedanib) Route of administration: oral Twice daily (to be swallowed unchewed with a glass of water of about 250 mL. If taken twice the dose interval should be of around 12 hours at the same times every day, usually in the morning and the evening after food intake).
  Continuous daily dosing until progression of disease or until criteria for interruption of treatment is met, no intake of placebo on days of paclitaxel and carboplatin administration.
  The maximum time on monotherapy is 2 years.
  Arms: placebo

SUMMARY:
Patients with extensive and bulky disease are often those whose initial surgery is delayed after 3 or 4 cycles of neo-adjuvant chemotherapy.

In that case, there is, indeed, some concern to administer bevacizumab during the chemotherapy surrounding the interval debulking surgery due to the long half life (14- 21 days) of this monoclonal antibody and the interference of anti angiogenic agents with wound healing.

Vargatef® (Nintedanib) might offer a better alternative to bevacizumab in the neo-adjuvant setting. Vargatef® (Nintedanib) has a much shorter half-life of 7 to 19 hours. Preliminary experience in cancer did not show a trend for increased incidence of fistula or bowel perforation. For more details please refer to the investigator drug brochure for Vargatef® (Nintedanib).

This trial will compare progression-free survival and surgical complications of 188 patients with FIGO stage IIIC/IV treated in first line with either neo-adjuvant chemotherapy (carboplatin & paclitaxel) and interval debulking surgery or the same treatment + Vargatef® (Nintedanib).

ELIGIBILITY:
Inclusion Criteria:

* First diagnosis of histological confirmed (cytology alone excluded) epithelial ovarian cancer, fallopian tube or primary peritoneal cancer. Histology should be obtained by laparoscopy (or by laparotomy),
* FIGO-Stages IIIC - IV,
* ECOG performance status < 2,
* Life expectancy of at least 6 months,
* Primary debulking surgery denied and maximum surgical effort of cytoreduction with the goal of no residual disease planned as interval debulking surgery,
* Interval between diagnosis and enrolment (informed consent) ≤ 8 weeks,
* Adequate hepatic, renal and bone marrow functions:

Platelets > 100 000 /μL, Hemoglobin > 9.0 g/dL, Absolute Neutrophil Count (ANC) > 1500/μL, Prothrombin time and/or partial thromboplastin time < 50% deviation from normal limits in the absence of therapeutic anticoagulation, Proteinuria < CTCAE grade 2, Total bilirubin ≤ upper limit of normal (ULN), ALT and/or AST ≤ 2.5 x ULN, Glomerular filtration rate >40 mL/min,

* Females, age 18 years or older,
* Patient has given written informed consent,

Exclusion Criteria:

* Histological diagnosis of malignant tumour of non-epithelial origin (e.g. germ cell tumour, malignant mixed mullerian tumour, sex cord-stromal tumour) of the ovary, the fallopian tube or peritoneum or borderline tumour of the ovary (tumour of low malignant potential),
* Non-healing wound, ulcer (intestinal tract, skin) or bone fracture,
* Clinical symptoms or signs of gastrointestinal obstruction,
* History of major thromboembolic event, defined as:

  * Pulmonary embolism (PE) within 6 months prior to enrolment,
  * Recurrent pulmonary embolism (history of at least 2 events),
* History of at least 2 unprovoked (without a transient or reversible risk factor) events of proximal deep venous thrombosis,
* Prior thrombosis or thromboembolic event in the presence of an inherited coagulopathy (including deficiency of antithrombin, deficiency of protein C or protein S, Factor V Leiden mutation, Prothrombin G20210A mutation),
* Patients with perioperative thrombosis including proximal deep vein thrombosis (DVT) or thrombosis of visceral vessels not associated with pulmonary embolism may be included in the trial if stable therapeutic anticoagulation is documented,
* Known inherited or acquired bleeding disorder,
* Significant cardiovascular diseases, including:

  * Hypertension not controlled by medical therapy,
  * Unstable angina within the past 6 months,
  * History of myocardial infarction within the past 6 months,
  * Congestive heart failure > NYHA II,
  * Clinically relevant cardiac arrhythmia
* Peripheral vascular disease Fontaine stage ≥3,
* Clinically relevant pericardial effusion (e.g. pericardial effusion with echocardiographic or clinical signs of haemodynamic impairment),
* History of a cerebral vascular accident, transient ischemic attack or subarachnoid hemorrhage within the past 6 months,
* Serious infections in particular if requiring systemic antibiotic (antimicrobial, antifungal) or antiviral therapy, including HIV-infection, hepatitis B and/or C infection,
* Poorly controlled diabetes mellitus or other contraindication to high dose corticosteroid therapy,
* Clinical symptoms of brain metastases and/or diagnosis of brain metastases on imaging,
* Pre-existing sensory or motor neuropathy CTCAE ≥ 2, except due to trauma,
* Gastrointestinal disorders or abnormalities that would interfere with absorption of the study drug,
* Other malignancy diagnosed within the past 5 years, except:

  * non-melanomatous skin cancer (if adequately treated),
  * cervical carcinoma in situ (if adequately treated),
  * carcinoma in situ of the breast (if adequately treated),
  * prior or synchronous endometrial cancer (if adequately treated), provided the following criteria are met:

    * Disease stage FIGO ≤ IB,
    * No more than superficial myometrial invasion,
    * Not poorly differentiated (less than grade 3, no papillary serous or clear cell histology),
* Prior systemic therapy for ovarian cancer (e.g. chemotherapy, monoclonal antibody therapy, oral targeted therapy, hormonal therapy),
* Prior radiotherapy to the abdomen or prior radiotherapy to an extra-abdominal target volume that would bear the risk of increased toxicity of chemotherapy,
* Hypersensitivity to Vargatef® (Nintedanib) and/or the excipients of the trial drugs,
* Serious illness or concomitant non-oncological disease such as neurologic, psychiatric or infectious disease, active ulcers (gastrointestinal tract, skin) or a laboratory abnormality that may increase the risk associated with study participation or study drug administration and in the judgment of the investigator would make the patient inappropriate for entry into the study,
* Patients with preserved reproductive capacity who are sexually active and unwilling to use a medically acceptable method of contraception (e.g. such as implants, injectables, combined oral contraceptives, some intrauterine devices or vasectomized partner) during the trial and for at least twelve months after end of active therapy,
* Pregnancy or breast feeding,
* Psychological, familial, sociological or geographical factors potentially hampering compliance with the study protocol and follow-up schedule,
* Active alcohol or drug abuse,
* Any contraindications for therapy with paclitaxel or carboplatin, e.g. a history of severe hypersensitivity reactions to paclitaxel or platinum-containing compounds and their excipients, or other drugs formulated with Polyoxyl 35 Castor Oil - ELP,
* Treatment with other investigational drugs or participation in another clinical trial testing a drug within the past four weeks before start of therapy or concomitantly with this trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2012-06; Primary Completion 2015-05 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Median Progression-free Survival (PFS) in each study arm | average of 18 months

SECONDARY OUTCOMES:
Response rate | 2 months after beginning of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Gwénaël Ferron, MD, Principal Investigator — Institut Claudius Régaud
Locations (36):
- France (36):
  - Centre Paul Papin, Angers
  - Institut Ste Catherine, Avignon
  - Clinique Tivoli, Bordeaux
  - Institut Bergonié, Bordeaux
  - Polyclinique Bordeaux Nord, Bordeaux
  - Centre François Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Hospitalier Alpes Leman, Contamine-sur-Arve
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - Centre Hospitalier de Dax, Dax
  - Centre Georges François Leclerc, Dijon
  - Centre Hospitalier Régional Universitaire de Lille - Hôpital Huriez, Lille
  - Centre Oscar Lambret, Lille
  - Centre Hospitalier Universitaire Dupuytren, Limoges
  - Centre Léon bérard, Lyon
  - ICM Val d'Aurelle, Montpellier
  - Centre Catherine de Sienne, Nantes
  - Hôpital Privé du Confluent S.A.S., Nantes
  - Centre Antoine Lacassagne, Nice
  - Centre Hospitalier Régional, Orléans
  - Hôpital Cochin, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Tenon, Paris
  - Institut Mutualiste Montsouris-Jourdan, Paris
  - Centre Hospitalier Lyon-sud, Pierre-Bénite
  - Milétrie - Centre Hospitalier Universitaire de Poitiers, Poitiers
  - Institut Jean Godinot, Reims
  - Centre Henri Becquerel, Rouen
  - Clinique Armoricaine de Radiologie, Saint-Brieuc
  - Hôpital René Huguenin, Saint-Cloud
  - ICO René Gauducheau, Saint-Herblain
  - Hôpital Civil, Strasbourg
  - Hôpitaux Du Leman, Thonon-les-Bains
  - Centre Claudius Régaud, Toulouse
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Gustave Roussy, Villejuif

REFERENCES:
- [Derived] Marchetti C, Ferron G, Colomban O, Giannarelli D, Blanc-Durand F, Scambia G, Just PA, Lorusso D, Pujade-Lauraine E, Ergasti R, Lortholary A, Sassu CM, Ray-Coquard I, Capomacchia FM, Combe P, Apostol AI, Zannoni GF, Carrot A, Malapelle U, Leary A, Fagotti A, You B. Predictors of Successful Neoadjuvant Chemotherapy and Interval Cytoreductive Surgery in Management of Ovarian Cancer. JCO Oncol Pract. 2025 Nov 24:OP2500469. doi: 10.1200/OP-25-00469. Online ahead of print. PMID 41284952
- [Derived] Azais H, Brochard C, Taly V, Benoit L, Ferron G, Ray-Coquard I, You B, Abadie-Lacourtoisie S, Lebreton C, Venat L, Louvet C, Favier L, Blonz C, Dohollou N, Malaurie E, Dubot C, Kurtz JE, Pujade-Lauraine E, Rouleau E, Leary A, Bats AS, Blons H, Laurent-Puig P. Prognostic value of circulating tumor DNA at diagnosis and its early decrease after one cycle of neoadjuvant chemotherapy for patients with advanced epithelial ovarian cancer. An ancillary analysis of the CHIVA phase II GINECO trial. Gynecol Oncol. 2025 Jan;192:145-154. doi: 10.1016/j.ygyno.2024.12.004. Epub 2024 Dec 12. PMID 39671779
- [Derived] Yaniz-Galende E, Zeng Q, Bejar-Grau JF, Klein C, Blanc-Durand F, Le Formal A, Pujade-Lauraine E, Chardin L, Edmond E, Marty V, Ray-Coquard I, Joly F, Ferron G, Pautier P, Berton-Rigaud D, Lortholary A, Dohollou N, Desauw C, Fabbro M, Malaurie E, Bonichon-Lamaichhane N, Bello Roufai D, Gantzer J, Rouleau E, Genestie C, Leary A. Spatial Profiling of Ovarian Carcinoma and Tumor Microenvironment Evolution under Neoadjuvant Chemotherapy. Clin Cancer Res. 2024 Jul 1;30(13):2790-2800. doi: 10.1158/1078-0432.CCR-23-3836. PMID 38669064
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961
- [Derived] Ferron G, De Rauglaudre G, Becourt S, Delanoy N, Joly F, Lortholary A, You B, Bouchaert P, Malaurie E, Gouy S, Kaminsky MC, Meunier J, Alexandre J, Berton D, Dohollou N, Dubot C, Floquet A, Favier L, Venat-Bouvet L, Fabbro M, Louvet C, Lotz JP, Abadie-Lacourtoisie S, Desauw C, Del Piano F, Leheurteur M, Bonichon-Lamichhane N, Rastkhah M, Follana P, Gantzer J, Ray-Coquard I, Pujade-Lauraine E. Neoadjuvant chemotherapy with or without nintedanib for advanced epithelial ovarian cancer: Lessons from the GINECO double-blind randomized phase II CHIVA trial. Gynecol Oncol. 2023 Mar;170:186-194. doi: 10.1016/j.ygyno.2023.01.008. Epub 2023 Jan 25. PMID 36706645
- [Derived] Aide N, Fauchille P, Coquan E, Ferron G, Combe P, Meunier J, Alexandre J, Berton D, Leary A, De Rauglaudre G, Bonichon N, Pujade Lauraine E, Joly F. Predicting tumor response and outcome of second-look surgery with 18F-FDG PET/CT: insights from the GINECO CHIVA phase II trial of neoadjuvant chemotherapy plus nintedanib in stage IIIc-IV FIGO ovarian cancer. Eur J Nucl Med Mol Imaging. 2021 Jun;48(6):1998-2008. doi: 10.1007/s00259-020-05092-3. Epub 2020 Nov 21. PMID 33221969
- [Derived] Robelin P, Tod M, Colomban O, Lachuer J, Ray-Coquard I, Rauglaudre G, Joly F, Chevalier-Place A, Combe P, Lortholary A, Hamizi S, Raban N, Ferron G, Meunier J, Berton-Rigaud D, Alexandre J, Kaminsky MC, Dubot C, Leary A, Malaurie E, You B. Comparative analysis of predictive values of the kinetics of 11 circulating miRNAs and of CA125 in ovarian cancer during first line treatment (a GINECO study). Gynecol Oncol. 2020 Oct;159(1):256-263. doi: 10.1016/j.ygyno.2020.07.021. Epub 2020 Jul 22. PMID 32712155